CLINICAL TRIAL: NCT01369381
Title: Intubation Mechanics of the Stable and Unstable Cervical Spine
Brief Title: Cervical Spine Biomechanics During Endotracheal Intubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Collaborators: National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH); Colorado State University (Other)
Responsible Party: Principal Investigator, Bradley J. Hindman, Professor, Department of Anesthesia, University of Iowa
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 201102721; R01EB012048 (NIH)
Record Dates: First submitted 2011-05-31; First posted 2011-06-08 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-08

CONDITIONS: Spinal Diseases; Other Biomechanical Lesions of Cervical Region; Tracheal Intubation Morbidity
Keywords: Cervical spine; Endotracheal intubation; Laryngoscope; Biomechanics
MeSH Terms: conditions — Spinal Diseases | interventions — Intubation, Intratracheal

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Airtraq laryngoscope (Experimental): The Airtraq is an alternative indirect laryngoscope that appears to cause less cervical spine motion during intubation that conventional direct laryngoscopy (Macintosh blade)
  Interventions: Procedure: Endotracheal intubation
- Macintosh laryngoscope (Active Comparator): This arm constitutes intubation with a conventional direct laryngoscopy with a Macintosh blade which has been shown to result in cervical spine extension, particularly in the upper cervical segments.
  Interventions: Procedure: Endotracheal intubation

INTERVENTIONS:
Procedure: Endotracheal intubation — Study patients undergo endotracheal intubation using both a conventional direct laryngoscope (Macintosh) and an alternative indirect laryngoscope (Airtraq). The order of intubation (Macintosh then Airtraq--or--Airtraq then Macintosh) is randomized.

SUMMARY:
Current methods for endotracheal intubation in the presence of cervical spine (c-spine) instability are not evidence-based. This is so because the relationships between the forces applied during intubation (by the laryngoscope) and the resulting c-spine movement have not yet been quantitatively characterized. As a result, with the current level of knowledge, it is not known, and it is not possible to predict, which types of c-spine instability have the greatest risk of cervical spinal cord injury with intubation. This shortcoming makes it impossible to know which intubation devices and techniques are likely to be safest in the presence of c-spine instability.

To address this critical lack of knowledge, the overarching purpose of the proposed research is to: 1) quantitatively relate c-spine movement that results from the forces applied to the peri-airway tissues during intubation (force-motion relationships), and 2) use these data to develop a mathematical model of the c-spine that will predict which types of c-spine instability result in the greatest amount of abnormal c-spine motion and associated spinal cord compression during intubation.

This clinical study will utilize laryngoscope blades that are instrumented with a high resolution pressure mapping system to make high-resolution measurements of the forces and pressures of intubation while making simultaneous measurements of c-spine motion. In this study, study subjects will be intubated using both a conventional (Macintosh) laryngoscope and an alternative (Airtraq) laryngoscope. By using two different laryngoscopes, we, the investigators, will introduce forces of differing magnitudes and distributions to peri-airway tissues. The Airtraq does not require a direct line of sight to visualize the vocal cords, and among the various new alternative laryngoscopes it is the only one that has been shown to result in 30-50% less cervical motion than a conventional (Macintosh) laryngoscope. Accordingly, we hypothesize 1) 30-50% less force will be applied with the Airtraq laryngoscope than with the conventional (Macintosh) laryngoscope and 2) 30-50% less c-spine motion will occur with the Airtraq. By studying (intubating) each subject twice, any differences in the c-spine force-motion relationships between devices will be due to the devices themselves. By studying each subject twice, we can account for (and eliminate) differences among study subjects in c-spine biomechanical properties.

ELIGIBILITY:
Inclusion Criteria:

* Patient Height: 5-feet, 0-inches to 6-feet, 0-inches
* Patient body mass index: less than 30 kg/m2
* Planned surgery requires use of C-arm fluoroscopy
* Planned surgery to take place at University of Iowa and requires general anesthesia and orotracheal intubation

Exclusion Criteria:

* The patient is a prisoner
* The patient is pregnant
* The patient is not competent to personally give consent
* Neurological signs and symptoms indicating cervical spinal cord myelopathy
* Cervical spine images demonstrating anatomic instability, traumatic injury, significant cervical stenosis, and/or spinal immobility
* Condition associated with cervical spine anatomic abnormalities such as Rheumatoid arthritis, Down Syndrome, Ankylosing spondylitis, Osteogenesis imperfecta
* Prior cervical spine surgery of any type
* History of difficult endotracheal intubation
* Currently symptomatic gastroesophageal reflux disease
* Currently symptomatic asthma or other reactive airway disease
* Any history of coronary artery disease
* Any history of cerebral aneurysm(s)
* History of vocal cord and/or glottic disease or dysfunction
* Contraindication to receiving 100% oxygen
* Systolic blood pressure greater than 180 mmHg
* Diastolic blood pressure greater than 100 mmHg
* American Society of Anesthesiologists Physical Status class of 4, 5, or 6
* Known allergy or other adverse response to study drugs: midazolam, lidocaine, fentanyl, propofol [eggs, soy beans], rocuronium, or sevoflurane.
* Mallampati oropharyngeal class of III or IV
* Thyromental distance less than 6.0 cm
* Sternomental distance less than 12.5 cm
* Maxillary incisors loss or in poor condition

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2011-12; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Cervical spine segmental intervertebral motion | Data collection takes place during two sequential endotracheal intubations (40-45 seconds), with follow-up assessments on postoperative days 1, 3, and 7.
  Lateral fluoroscopy is used to measure cervical spine motion during endotracheal intubation.

SECONDARY OUTCOMES:
Laryngoscope blade force distribution | Data collection takes place during two sequential endotracheal intubations (40-45 seconds), with follow-up assessments on postoperative days 1, 3, and 7.
  "Pressure-mat" technology is used to measure spacially distributed forces applied by the laryngoscope blade during endotracheal intubation.
Glottic visualization | Data collection takes place during two sequential endotracheal intubations (40-45 seconds), with follow-up assessments on postoperative days 1, 3, and 7.
  An image of the glottis during intubation is obtained for off-line measurement of the percentage of glottic opening as seen by the laryngoscopist.

CONTACTS AND LOCATIONS:
Overall Officials: Bradley J Hindman, M.D., Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

REFERENCES:
- [Background] LeGrand SA, Hindman BJ, Dexter F, Weeks JB, Todd MM. Craniocervical motion during direct laryngoscopy and orotracheal intubation with the Macintosh and Miller blades: an in vivo cinefluoroscopic study. Anesthesiology. 2007 Dec;107(6):884-91. doi: 10.1097/01.anes.0000291461.62404.46. PMID 18043056
- [Background] Santoni BG, Hindman BJ, Puttlitz CM, Weeks JB, Johnson N, Maktabi MA, Todd MM. Manual in-line stabilization increases pressures applied by the laryngoscope blade during direct laryngoscopy and orotracheal intubation. Anesthesiology. 2009 Jan;110(1):24-31. doi: 10.1097/ALN.0b013e318190b556. PMID 19104166
- [Background] Hindman BJ, Palecek JP, Posner KL, Traynelis VC, Lee LA, Sawin PD, Tredway TL, Todd MM, Domino KB. Cervical spinal cord, root, and bony spine injuries: a closed claims analysis. Anesthesiology. 2011 Apr;114(4):782-95. doi: 10.1097/ALN.0b013e3182104859. PMID 21326090
- [Background] Hirabayashi Y, Fujita A, Seo N, Sugimoto H. A comparison of cervical spine movement during laryngoscopy using the Airtraq or Macintosh laryngoscopes. Anaesthesia. 2008 Jun;63(6):635-40. doi: 10.1111/j.1365-2044.2008.05480.x. PMID 18477276
- [Background] Turkstra TP, Pelz DM, Jones PM. Cervical spine motion: a fluoroscopic comparison of the AirTraq Laryngoscope versus the Macintosh laryngoscope. Anesthesiology. 2009 Jul;111(1):97-101. doi: 10.1097/ALN.0b013e3181a8649f. PMID 19512871
- [Derived] Hindman BJ, Dexter F, Gadomski BC, Puttlitz CM. Relationship Between Glottic View and Intubation Force During Macintosh and Airtraq Laryngoscopy and Intubation. Anesth Analg. 2022 Oct 1;135(4):815-819. doi: 10.1213/ANE.0000000000006082. Epub 2022 May 13. PMID 35551148